CLINICAL TRIAL: NCT07088731
Title: A Prospective, Single-Center, Randomized Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Nab-Paclitaxel Combined With Cisplatin and Sintilimab in Neoadjuvant Treatment of Locally Advanced Cervical Cancer
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Nab-Paclitaxel Combined With Cisplatin and Sintilimab in Neoadjuvant Treatment of Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, GUANG WEN YUAN, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25/275-5221
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cervical Carcinoma
Keywords: locally advanced; neoadjuvent chemotherapy; neoadjuvent immunotherapy; CCRT
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — sintilimab; 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvent arm (Experimental)
  Interventions: Drug: Sintilimab
- CCRT arm (Active Comparator)
  Interventions: Radiation: Concurrent chemo-radiotherapy

INTERVENTIONS:
Drug: Sintilimab — neoadjuvent chemotherapy plus sintilimab for 2 cycles followed by radical surgery
  Other Names: Nab-paclitaxel; cisplatin
  Arms: neoadjuvent arm
Radiation: Concurrent chemo-radiotherapy — EBRT+BT+cisplatin
  Arms: CCRT arm

SUMMARY:
For locally advanced cervical cancer, there are two main treatment options:

One is radical chemoradiotherapy (a combination of radiotherapy and chemotherapy aimed at curing the disease).

The other is having neoadjuvant treatment first (treatment given before the main surgery to shrink the tumor) followed by radical surgery.

So far, there's no clear answer on which of these two options is better. In general, cervical cancer responds well to immunotherapy. But we still don't know for sure if adding immunotherapy to neoadjuvant chemotherapy can improve the treatment effect for locally advanced cervical cancer, or even make it better than radical chemoradiotherapy.

This study aims to compare the effects of two approaches: radical chemoradiotherapy versus neoadjuvant chemotherapy plus immunotherapy followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and ≤ 70 years;
* Cervical cancer with pathological types being squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma;
* Staged IB3 or IIA2 according to the FIGO 2018 staging system, as assessed by the investigator;
* ECOG performance status of 0-2, or KPS score ≥ 70;
* Expected survival time of more than 3 months;
* Having at least one measurable lesion in accordance with RECIST 1.1;
* Laboratory test results meeting the following criteria without drug intervention:

  1. Hemoglobin ≥ 90 g/dl, neutrophil count ≥ 1.5 × 10⁹/L, platelet count ≥ 100 × 10⁹/L;
  2. Creatinine ≤ 1.5 times the upper limit of normal range;
  3. Total bilirubin, alanine transaminase (ALT), and aspartate transaminase (AST) < 2 times the upper limit of normal;
* Postmenopausal, or reproductive-aged women who meet all the following conditions: non-lactating, not pregnant, and able to use effective contraceptive measures during the study treatment period;
* Voluntarily participating in this study and signing the informed consent form.

Exclusion Criteria:

* Participated in other clinical trials within 30 days before receiving the first dose of chemotherapy drugs or during the treatment period.
* Previously received any other anti-tumor treatment for cervical cancer.
* Non-HPV-related cervical cancer.
* Needing to receive other anti-tumor treatments during the study treatment period.
* Patients with known allergies to the active ingredients of the study drugs or their excipients.
* Diagnosed with other malignant tumors in the past 5 years (except those judged to be cured by the investigator).
* Active infections requiring systemic treatment.
* Positive for human immunodeficiency virus (HIV) antibody.
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody.
* Peripheral neuropathy with a grade of ≥ 2 according to the NCI-CTCAE (Version 5.0).
* Concurrent diseases or abnormal test results that interfere with the subject's ability to receive anti-tumor treatment as judged by the investigator, such as the estimated inability of the subject to tolerate at least 2 cycles of neoadjuvant chemotherapy plus surgery or concurrent chemoradiotherapy, etc.

Participation in this study is deemed not conducive to the maximum benefit of the subject as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
2-year Progression-Free Survival Rate | From enrollment to the end of treatment at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecological Oncology, Beijing, China